CLINICAL TRIAL: NCT07392099
Title: Comparison of the Efficacy of an Empowered Relief Single-Session Versus Standard Care for Reducing Postoperative Pain Following Elective Orthopedic Surgery: A Randomized Controlled Trial
Acronym: ER-CHUS -Ortho
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Estrie University Integrated Health and Social Services Center - University Hospital of Sherbrooke (Other)
Responsible Party: Principal Investigator, Junie Carrière, Assistant Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CÉRCIUSSSEstrieCHUS_2025-5666
Record Dates: First submitted 2025-08-25; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: Postoperative Pain; Elective Orthopedic Surgery; chronic pain; behavioral health
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Clinical trial randomizing to one of two groups: (1) standard care; and (2) single-session pain relief skills intervention for chronic pain (Empowered Relief)
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and research staff will know arm assignment. Co-investigators, project statisticians, and the protocol director at each study site will remain blinded until final assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowered Relief (ER) (Experimental): Behavioral: Empowered Relief A certified instructor delivers 1 session of pain relief skills intervention (Empowered Relief) to groups of patients who were randomized to this treatment arm.The ER session will be done between 4 to 8 weeks before the surgery. All treatment sessions will be conducted in person, in a meeting room of the CIUSSS de l'Estrie-CHUS
  Interventions: Behavioral: Empowered Relief (ER) consists of a single-session, 2-hour group class.
- Waitlist Control (WLC) (No Intervention): Participants randomized to the waitlist control arm will be instructed to continue with their usual medical care.

INTERVENTIONS:
Behavioral: Empowered Relief (ER) consists of a single-session, 2-hour group class. — ER is rooted in cognitive behavioral theory and incorporates pain education, self-regulatory skills and mindfulness principle
  Arms: Empowered Relief (ER)

SUMMARY:
The purpose of this study is to evaluate the efficacy and acceptability of the French-Canadian version of ER compared to standard care in reducing postoperative pain and improving recovery outcomes at 6-week and 3-month follow-ups after elective orthopedic surgery.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a pragmatic clinical trial comparing the effectiveness and acceptability of two postoperative pain management approaches following elective orthopedic surgery:

1. Empowered Relief (ER): A single-session, 2-hour intervention based on cognitive behavioral therapy (CBT) principles, designed to teach patients pain self-management strategies.
2. Standard Care: Usual postoperative care without additional psychological intervention.

The investigators aim to determine which approach is more effective and acceptable for patients in managing postoperative pain. Ultimately, this research aims to provide a low-cost, low-risk, widely accessible, and feasible intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pain >4/10 for >3 months related to the surgical indication
* French fluency
* Ability to adhere to and complete study protocol
* Males and females, 18+

Exclusion Criteria:

* Participated in another project that may cause bias in the study results
* Pain related to cancer
* Cognitive impairment, non-French speaking, or factors that would preclude comprehension of material or full participation in ER
* Previous participation in ER

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity and Interference | 6-weeks post-surgery
  The Brief Pain Inventory-short form measures both the intensity of pain and the interference of pain in various aspects of the patient's life. Patients rate their pain at its "worst," "least," "average," and "now" (current pain) over the past 24 hours. Ratings are provided on a scale from 0 to 10, where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine." Patients also assess how pain has interfered with seven aspects of their daily life: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
Pain Intensity and Interference | 3-months post-surgery
  The Brief Pain Inventory-short form measures both the intensity of pain and the interference of pain in various aspects of the patient's life. Patients rate their pain at its "worst," "least," "average," and "now" (current pain) over the past 24 hours. Ratings are provided on a scale from 0 to 10, where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine." Patients also assess how pain has interfered with seven aspects of their daily life: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life.
Treatment Acceptability | Less than 7 days Post ER session
  Acceptability of the ER session will be assessed with the Acceptability Home-based questionnaire, a 8-item measure with a total score ranging from 0-48 with higher scores indicative of more acceptability.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | 6-weeks post-surgery
  Pain Catastrophizing Scale is a 13-item measure with a total score ranging from 0-52 with higher scores indicative of more catastrophizing.
Pain Catastrophizing Scale | 3-months post-surgery
  Pain Catastrophizing Scale is a 13-item measure with a total score ranging from 0-52 with higher scores indicative of more catastrophizing.
Pain Self-Efficacy Questionnaire (PSEQ) | 6-weeks post-surgery
  The 10 item Pain Self-Efficacy Questionnaire (PSEQ) assesses self-efficacy using à 0 = "Not confident at all" to 6= "Completely confident" scale. Higher scores suggest a greater self-efficacy.
Pain Self-Efficacy Questionnaire (PSEQ) | 3-months post-surgery
  The 10 item Pain Self-Efficacy Questionnaire (PSEQ) assesses self-efficacy using à 0 = "Not confident at all" to 6= "Completely confident" scale. Higher scores suggest a greater self-efficacy.
General Self-Efficacy - Short Form 4a | 6-weeks post-surgery
  Compare treatment groups for self-efficacy using the PROMIS 4-item PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Self-Efficacy - Lower scores indicate lower levels of Self-Efficacy.
General Self-Efficacy - Short Form 4a | 3-months post-surgery
  Compare treatment groups for self-efficacy using the PROMIS 4-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Self-Efficacy - Lower scores indicate lower levels of Self-Efficacy.
PROMIS Short Form v1.0 - Depression - 8a | 6-weeks post-surgery
  Compare treatment groups for depression using the PROMIS 8-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Depression - Lower scores indicate lower levels of Depression.
PROMIS Short Form v1.0 - Depression - 8a | 3-months post-surgery
  Compare treatment groups for depression using the PROMIS 8-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Depression - Lower scores indicate lower levels of Depression.
PROMIS Short Form v1.0 - Anxiety - 8a | 6-weeks post-surgery
  Compare treatment groups for anxiety using the PROMIS 8-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Anxiety- Lower scores indicate lower levels of Anxiety.
PROMIS Short Form v1.0 - Anxiety - 8a | 3-months post-surgery
  Compare treatment groups for anxiety using the PROMIS 8-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Anxiety- Lower scores indicate lower levels of Anxiety.
PROMIS Short Form v1.0 - Sleep Disturbance 4a | 6-weeks post-surgery
  Compare treatment groups for sleep disturbance using the PROMIS 4-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Sleep disturbance - Lower scores indicate lower levels of Sleep disturbance.
PROMIS Short Form v1.0 - Sleep Disturbance 4a | 3-months post-surgery
  Compare treatment groups for sleep disturbance using the PROMIS 4-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Sleep disturbance - Lower scores indicate lower levels of Sleep disturbance.
PROMIS Short Form v2.0 - Social Isolation 4a | 6-weeks post-surgery
  Compare treatment groups for social isolation using the PROMIS 4-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Social isolation - Lower scores indicate lower levels of Social isolation.
PROMIS Short Form v2.0 - Social Isolation 4a | 3-months post-surgery
  Compare treatment groups for social isolation using the PROMIS 4-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Social isolation - Lower scores indicate lower levels of Social isolation.
PROMIS Short Form v1.0 - Fatigue 4a | 6-weeks post-surgery
  Compare treatment groups for fatigue using the PROMIS 4-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Fatigue - Lower scores indicate lower levels of Fatigue.
PROMIS Short Form v1.0 - Fatigue 4a | 3-months post-surgery
  Compare treatment groups for fatigue using the PROMIS 4-item. PROMIS instruments are normed on the US population and are reported using t-scores with a mean of 50 and a standard deviation of 10.
  Higher scores indicate higher levels of Fatigue - Lower scores indicate lower levels of Fatigue.
Short Assessment of Patient Satisfaction (SAPS) | 3-months post-surgery
  The Short Assessment of Patient Satisfaction (SAPS) assesses patients' satisfaction regarding their health care with 7 items using a 4 likert scale from "very satisfied" to "very unsatisfied"

OTHER OUTCOMES:
Pain medication | Baseline
  Pain medication use will be assessed using a self-report medication questionnaire asking participants which medications they have used to relieve pain in the past 2 weeks. Medication categories include:
  Acetaminophen, Non-steroidal anti-inflammatory drugs (NSAIDs), Muscle relaxants, Opioid/narcotic analgesics, Neuropathic pain medications (e.g., gabapentin, pregabalin), Antidepressants used for pain, Cannabis and Other (specified by participant). For each category, participants indicate frequency of use: As needed (occasionally), Regularly, Used previously but stopped.
Pain medication | 6-weeks post-surgery
  Pain medication use will be assessed using a self-report medication questionnaire asking participants which medications they have used to relieve pain in the past 2 weeks. Medication categories include:
  Acetaminophen, Non-steroidal anti-inflammatory drugs (NSAIDs), Muscle relaxants, Opioid/narcotic analgesics, Neuropathic pain medications (e.g., gabapentin, pregabalin), Antidepressants used for pain, Cannabis and Other (specified by participant). For each category, participants indicate frequency of use: As needed (occasionally), Regularly, Used previously but stopped.
Pain medication | 3-months post-surgery
  Pain medication use will be assessed using a self-report medication questionnaire asking participants which medications they have used to relieve pain in the past 2 weeks. Medication categories include:
  Acetaminophen, Non-steroidal anti-inflammatory drugs (NSAIDs), Muscle relaxants, Opioid/narcotic analgesics, Neuropathic pain medications (e.g., gabapentin, pregabalin), Antidepressants used for pain, Cannabis and Other (specified by participant). For each category, participants indicate frequency of use: As needed (occasionally), Regularly, Used previously but stopped.
Pain management method | 6-weeks post-surgery
  Use of non-pharmacological pain management approaches will be assessed using a self-report questionnaire asking participants which non-medication resources they consulted or used to relieve pain during the past month. Categories include: Physiotherapy, Occupational therapy, Massage therapy, Psychology services, Self-care strategies (e.g., ice, heat, self-massage), and Other (specified by participant). Participants will indicate frequency of use for each category: 1-2 times, 3-10 times, More than 10 times.
Pain management method | 3-months post-surgery
  Use of non-pharmacological pain management approaches will be assessed using a self-report questionnaire asking participants which non-medication resources they consulted or used to relieve pain during the past month. Categories include: Physiotherapy, Occupational therapy, Massage therapy, Psychology services, Self-care strategies (e.g., ice, heat, self-massage), and Other (specified by participant). Participants will indicate frequency of use for each category: 1-2 times, 3-10 times, More than 10 times.

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSSE de l'Estrie CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No